CLINICAL TRIAL: NCT01931644
Title: A Multi-Site Tissue Repository Providing Annotated Biospecimens for Approved Investigator-Directed Biomedical Research Initiatives
Brief Title: At-Home Research Study for Patients With Autoimmune, Inflammatory, Genetic, Hematological, Infectious, Neurological, CNS, Oncological, Respiratory, Metabolic Conditions
Status: Completed | Type: Observational
Sponsor: Sanguine Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-BB-01
Record Dates: First submitted 2013-08-23; First posted 2013-08-29 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: All Diagnosed Health Conditions; ADD/ADHD; Alopecia Areata; Ankylosing Spondylitis; Asthma; Atopic Dermatitis Eczema; Beta Thalassemia; Bipolar Disorder; Breast Cancer; Celiac Disease; Cervical Cancer; Chronic Inflammatory Demyelinating Polyneuropathy; Chronic Kidney Diseases; Chronic Obstructive Pulmonary Disease; Colon Cancer; Colorectal Cancer; Crohn's Disease; Cystic Fibrosis; Depression; Diabetes Mellitus; Duchenne Muscular Dystrophy; Endometriosis; Epilepsy; Facioscapulohumeral Muscular Dystrophy; G6PD Deficiency; General Anxiety Disorder; Hepatitis B; Hereditary Hemorrhagic Telangiectasia; HIV/AIDS; Human Papilloma Virus; Huntington's Disease; Idiopathic Thrombocytopenic Purpura; Insomnia; Kidney Cancer; Leukemia; Lung Cancer; Lupus Nephritis; Lymphoma; Melanoma; Multiple Myeloma; Multiple Sclerosis; Myositis; Myotonic Dystrophy; Ovarian Cancer; Pancreatic Cancer; Parkinson's Disease; Polycystic Kidney Diseases; Prostate Cancer; Psoriasis; Psoriatic Arthritis; Rosacea; Scleroderma; Sickle Cell Anemia; Sickle Cell Trait; Sjogren's Syndrome; Skin Cancer; Spinal Muscular Atrophy; Systemic Lupus Erythematosus; Thrombotic Thrombocytopenic Purpura; Trisomy 21; Ulcerative Colitis
Keywords: ADD/ADHD; Alopecia Areata; Ankylosing Spondylitis; Asthma; Atopic Dermatitis Eczema; Beta Thalassemia; Bipolar Disorder; Breast Cancer; Celiac Disease; Cervical Cancer; Chronic Inflammatory Demyelinating Polyneuropathy; Chronic Kidney Diseases; Chronic Obstructive Pulmonary Disease; Colon Cancer; Colorectal Cancer; Crohn's Disease; Cystic Fibrosis; Depression; Diabete Mellitus; Duchenne Muscular Dystrophy; Endometriosis; Epilepsy; Facioscapulohumeral Muscular Dystrophy; G6PD Deficiency; General Anxiety Disorder; Hepatitis B; Hereditary Hemorrhagic Telangiectasia; HIV/AIDS; Human Papilloma Virus; Huntington's Disease; Idiopathic Thrombocytopenic Purpura; Insomnia; Kidney Cancer; Leukemia; Lung Cancer; Lupus Nephritis; Lymphoma; Melanoma; Multiple Myeloma; Multiple Sclerosis; Myositis; Myotonic Dystrophy; Ovarian Cancer; Pancreatic Cancer; Parkinson's Disease; Polycystic Kidney Diseases; Prostate Cancer; Psoriasis; Psoriatic Arthritis; Rosacea; Scleroderma; Sickle Cell Anemia; Sickle Cell Disease; Sickle Cell Trait; Sjogren's Syndrome; Skin Cancer; Spinal Muscular Atrophy; Systemic Lupus Erythematosus; Thrombotic Thrombocytopenic Purpura; Trisomy 21; Ulcerative Colitis
MeSH Terms: conditions — Alopecia Areata; Spondylitis, Ankylosing; Asthma; beta-Thalassemia; Bipolar Disorder; Breast Neoplasms; Celiac Disease; Uterine Cervical Neoplasms; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Renal Insufficiency, Chronic; Pulmonary Disease, Chronic Obstructive; Colonic Neoplasms; Colorectal Neoplasms; Crohn Disease; Cystic Fibrosis; Depression; Diabetes Mellitus; Muscular Dystrophy, Duchenne; Endometriosis; Epilepsy; Muscular Dystrophy, Facioscapulohumeral; Glucosephosphate Dehydrogenase Deficiency; Generalized Anxiety Disorder; Hepatitis B; Telangiectasia, Hereditary Hemorrhagic; Acquired Immunodeficiency Syndrome; Huntington Disease; Purpura, Thrombocytopenic, Idiopathic; Sleep Initiation and Maintenance Disorders; Kidney Neoplasms; Leukemia; Lung Neoplasms; Lupus Nephritis; Lymphoma; Melanoma; Multiple Myeloma; Multiple Sclerosis; Myositis; Myotonic Dystrophy; Ovarian Neoplasms; Pancreatic Neoplasms; Parkinson Disease; Polycystic Kidney Diseases; Prostatic Neoplasms; Psoriasis; Arthritis, Psoriatic; Rosacea; Scleroderma, Diffuse; Anemia, Sickle Cell; Sickle Cell Trait; Sjogren's Syndrome; Skin Neoplasms; Muscular Atrophy, Spinal; Lupus Erythematosus, Systemic; Purpura, Thrombotic Thrombocytopenic; Down Syndrome; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, PBMC, RNA, DNA, saliva, stool, hair, skin, CSF, synovial fuid, tumor tissue, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Health Condition: Collect blood and other optional biospecimens from participants with a diagnosed health condition
- Healthy Control: Collect blood and other optional biospecimens from participants that have not been diagnosed with a health condition

SUMMARY:
We are the missing link in clinical trials, connecting patients and researchers seamlessly and conveniently using a mobile health platform to advance medical research. We make it easy for patients to contribute to research for medical conditions that matter most to them, regardless of their location or ability to travel.

DETAILED DESCRIPTION:
This study will collect blood and other optionally donated tissue samples from people with all different types of health conditions, as well as healthy control samples, in order to provide biomedical researchers with quality biospecimens that are necessary in translating basic science research into clinically relevant information and technology.

ELIGIBILITY:
Inclusion Criteria:

* All adults 18-100 years old
* Able to provide proof of diagnosis
* Live in USA

Exclusion Criteria:

* Younger than 18 years old
* Receipt of blood products within 30 days of study blood collection
* Receipt of investigational drug within 30 days of study blood collection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosed with a health condition
Sampling Method: Probability Sample
Enrollment: 17667 (Actual)
Dates: Start 2013-07; Primary Completion 2024-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Biospecimen & Clinical Data Collection | 10 years
  To collect enough biospecimens and associated clinical data to allow researchers to come to statistically relevant scientific results

CONTACTS AND LOCATIONS:
Overall Officials: Houman Hemmati, MD, Principal Investigator — Sanguine Biosciences
Locations (1):
- Sanguine Biosciences, Los Angeles, California, United States